CLINICAL TRIAL: NCT03588156
Title: Single-dose Tolerability Study of Benapenem for Injection in Phase I Clinical Healthy Subjects
Brief Title: Single-dose PK Study of Benapenem In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5081-CPK-1001
Record Dates: First submitted 2018-05-16; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-05

CONDITIONS: Healthy Subject
Keywords: Healthy Subject; PK Study; Tolerability; Safety Evaluation
MeSH Terms: interventions — benapenem

STUDY DESIGN:
Intervention Model Description: 11 dose groups within 62.5 mg ~ 4000 mg for single-dose tolerability study to carried out from low-dose group to high-dose group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benapenem (Experimental): Investigatial Product: Benapenem: 11 group : 62.5mg one dose; 125mg one dose;250mg one dose;500mg one dose 30min infusion;500mg one dose 60min infusion ;1000mg one dose 30min infusion; 1000mg one dose 60min infusion 2000mg one dose 30min infusion;2000mg one dose 60min infusion;3000mg one dose 60min infusion;4000mg one dose 60min infusion
  Interventions: Drug: Benapenem
- Placebo (Placebo Comparator): Placebo control 11 group : 62.5mg one dose;125mg one dose;250mg one dose;500mg one dose 30min infusion;500mg one dose 60min infusion ;1000mg one dose 30min infusion; 1000mg one dose 60min infusion 2000mg one dose 30min infusion;2000mg one dose 60min infusion;3000mg one dose 60min infusion;4000mg one dose 60min infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benapenem — Dose-escalation For 11 level dose groups A1 ~ A11(each 62.5mg/kg, 125mg/kg, 250mg/kg, 500mg/kg, 1000mg/kg 60min infusion, 1000mg/kg 30min infusion, 2000mg/kg 60 min infusion, 2000mg/kg 30min infusion, 3000mg/kg, 4000mg/kg), 10 subjects (8 for the study drug and 2 for placebo) are randomized to each dose group
  Other Names: 5081
  Arms: Benapenem
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To design 11 dose groups within 62.5 mg ~ 4000 mg for single-dose tolerability study. A single-center, randomized, blinded, placebo-controlled, dose escalation trial design is adopted. 8 subjects each in 62.5 mg, 125 mg, 3000 mg and 4000 mg dose groups, 10 subjects each in other groups, including 2 placebo-controlled subjects. To be carried out from low-dose group to high-dose group. The next dose group can be studied only when the observation of the previous dose group is completed and it is confirmed that the drug is safely tolerated. The test should be stopped in case of serious adverse reactions, or when more subjects experience adverse reactions and have reached termination criteria of the trial, even if the maximum dose has not been reached.

Infusion time is planned to be 30 min in 62.5 mg, 125 mg and 250 mg ; two infusion time, 30 min and 60 min, in 500 mg, 1000 mg and 2000 mg groups. If subjects can tolerate 60-min infusion, the same dose group at infusion time of 30 min is added. The 3000 mg and 4000 mg dose groups only receive 60-min infusion for investigation of tolerability.

DETAILED DESCRIPTION:
It is planned to design 11 dose groups within 62.5 mg ~ 4000 mg for single-dose tolerability study. A single-center, randomized, blinded, placebo-controlled, dose escalation trial design is adopted. There are 8 subjects each in 62.5 mg, 125 mg, 3000 mg and 4000 mg dose groups, and 10 subjects each in other groups. Each group consists of half males and half females, including 2 placebo-controlled subjects (1 male and 1 female). The trial is carried out from low-dose group to high-dose group. Each subject only receives one dose of test drug, which is dissolved in 100 mL of 0.9% NS, intravenous drip. During the trial, the adverse events of subjects should be closely followed. The next dose group can be studied only when the observation of the previous dose group is completed and it is confirmed that the drug is safely tolerated. The test should be stopped in case of serious adverse reactions, or when more subjects experience adverse reactions and have reached termination criteria of the trial, even if the maximum dose has not been reached.

In order to investigate possible effect of infusion rate on the tolerability and to ensure the safety of subjects, the infusion time is planned to be 30 min in 62.5 mg, 125 mg and 250 mg low-dose groups; two infusion time, 30 min and 60 min, in 500 mg, 1000 mg and 2000 mg groups. Under the circumstance that subjects can tolerate 60-min infusion, the same dose group at infusion time of 30 min is added to investigate the possible effect of infusion rate on the tolerability. The 3000 mg and 4000 mg dose groups only receive 60-min infusion for investigation of tolerability.

ELIGIBILITY:
Inclusion Criteria:

* 1) Male or female healthy subjects, aged 18~45;
* 2) Body weight ≥ 50 kg and body mass index 19.0~24.0 kg/m2;
* 3) Prior to the test, physical examination, blood routine, urine routine, liver and kidney functions, and related examinations normal, or mild abnormalities in indicators while without clinical significance as indicated by the investigator;
* 4)Normal or mild abnormalities without clinical significance in the standard 12-lead ECG;
* 5)Signing informed consent form

Exclusion Criteria:

* 1) Regular smoking, alcohol abuse, and drug abuse;
* 2)Use of drugs known damage to an organ within three months;
* 3)History of specific allergies, or history of drug allergy, especially those allergic to lactams and excipients of test drug;
* 4)Febrile illnesses within three days before the screening;
* 5)Patients with mental illness or psychotic disorder in the past;
* 6)Past mental and nervous system diseases (epilepsy, stroke, cerebrovascular disorder, etc.), gastrointestinal disorder (such as stomach ulcers, gastritis, etc.) or disorder of other systems (such as cardiovascular, respiratory, hematological, or endocrine system, etc.) diseases or medical history.
* 7)Habitually taking any medication, including traditional Chinese medicine;
* 8)Having taken any medication that may affect test results within two weeks before the screening, such as antibiotics, NSAIDs, aluminum- or magnesium-containing antacids, diuretics, anticoagulants, central nervous system depressants, and any drug that may affect the drug absorption;
* 9)Having participated in other investigational drug trial in the preceding three months;
* 10)Blood donation for 360 ml or more within three months before the screening;
* 11)Heart rate < 50 bpm or > 100 bpm;
* 12)Systolic blood pressure<90mmHg or ≥ 140mmHg, diastolic blood pressure ≥ 90 mmHg or < 60 mmHg;
* 13)Women who are pregnant or breastfeeding, or who may be pregnant without adopting acceptable contraception, or who have a positive result in serum pregnancy test;
* 14)Women who are planning to become pregnant within 6 months, or male subjects who are planning to make his spouse pregnant within 6 months;
* 15)HBsAg, HCV antibody, HIV antibody, and Treponema pallidum antibody positive;
* 16)Urine drug-of-abuse testing positive;
* 17)Any other factor that makes the subject not suitable for the trial as indicated by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2015-09-17 (Actual); Study Completion 2015-09-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically significant findings in vital signs | Change from Baseline at Day1, Day2, Day4 after dosing
  Vitals signs such as systolic and diastolic blood pressure, heart rate, and pulse rate will be measured in a semi-supine position after 5 minutes of rest.
Number of subjects with clinically significant findings in laboratory parameters | Change from Baseline at Day1, Day2, Day4 after dosing
  Hematology and clinical chemistry and Urine Routine abnormalities will be monitored
Number of subjects with clinically significant 12-lead ECGs | Change from Baseline at Day1, Day2, Day4 after dosing
  Single 12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals

SECONDARY OUTCOMES:
AUC(0-24) of Benapenem | In each group: Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24hour after dosing
  AUC(0-24) is the area under the curve from time 0 to 24 hour
Maximum observed plasma concentration (Cmax) of Benepenem | In each group: Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24hour after dosing
Time to maximum observed plasma concentration (tmax) of Benapenem | In each group: Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24hour after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhu, Doctor, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data

REFERENCES:
- [Derived] Zhao CY, Lv Y, Zhu Y, Wei MJ, Liu MY, Ji XW, Kang ZS, Xia YH, Tian JH, Ma Y, Liu Y. A First-in-Human Safety, Tolerability, and Pharmacokinetics Study of Benapenem in Healthy Chinese Volunteers. Antimicrob Agents Chemother. 2019 Feb 26;63(3):e02188-18. doi: 10.1128/AAC.02188-18. Print 2019 Mar. PMID 30617093